CLINICAL TRIAL: NCT04221152
Title: A Multicenter, Open-label, Single-arm, Extension Study With Regard to the Safety and Efficacy of Empagliflozin in Patients With Refractory Diabetes Mellitus With Insulin Resistance (EMPIRE-02)
Brief Title: A Extension Study of Empagliflozin in Patients With Refractory Diabetes Mellitus With Insulin Resistance ( EMPIRE-02 )
Acronym: EMPIRE-02
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kobe University (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Wataru Ogawa, Professor, Division of Diabetes and Endocrinology, Kobe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190020
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Insulin Resistance - Type A; Insulin Resistance - Type B; Lipoatrophic Diabetes Mellitus; Insulin Resistance Syndrome
Keywords: insulin resistance; refractory diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Resistant, with Acanthosis Nigricans; Diabetes Mellitus, Lipoatrophic; Metabolic Syndrome; Insulin Resistance; Diabetes Mellitus | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of empagliflozin (Experimental): The study treatment shall be started from the next day of the Week 24 visit of the EMPIRE-01 study after enrollment. The investigational drug shall be administered at the same dosage as that of the empagliflozin tablet administered from Week 12 to Week 24 of the treatment period in the EMPIRE-01 study.
  The administration is oral administration with water once daily before or after breakfast.
  Interventions: Drug: Empagliflozin Tablets

INTERVENTIONS:
Drug: Empagliflozin Tablets — The administration is oral administration with water before or after breakfast.
  Other Names: BI10773

SUMMARY:
A multicenter, open-label, single-arm, extension study with regard to the safety and efficacy of empagliflozin in patients with refractory diabetes mellitus with insulin resistance.

DETAILED DESCRIPTION:
To determine the safety and efficacy of oral administration of empagliflozin 10 mg or 25 mg once daily for 28 weeks (52 weeks of the EMPIRE-01 study) in subjects who participated in the EMPIRE-01 study, which was conducted on refractory diabetes mellitus patients with insulin resistance (insulin resistance syndrome, lipoatrophic diabetes mellitus) in a multicenter, open-label, single-arm, extension study.

ELIGIBILITY:
Inclusion Criteria:

1. A patient who completed the preceding EMPIRE-01 study and does not meet any discontinuation criteria
2. A patient who has received sufficient explanation with regard to information such as the objectives and details of this study, expected drug efficacy/pharmacological action and risks, and has given written consent by her/himself

Exclusion Criteria:

1. A patient with a medical history of acute coronary syndrome (including non-ST-elevation myocardial infarction, ST-elevation myocardial infarction and unstable angina pectoris), stroke or transient ischemic attack (TIA) within 3 months before obtaining consent
2. A patient with suspected hepatic dysfunction that either of serum ALT, AST or alkaline phosphatase is exceeding 3-fold of upper limit of normal range prior to starting extension study treatment (Day 0)
3. A patient who is receiving a systemic steroid at the time of consent (except for type B)
4. A patient whose thyroid hormone product dose has been changed within 6 weeks before obtaining consent
5. A patient with unstable endocrine diseases other than diabetes mellitus
6. A patient with hemolysis or blood diseases that destabilize erythrocytic cells and other various disorders (e.g., malaria, babesiosis, hemolytic anemia)
7. A premenopausal female patient (the latest menstruation was within 1 year before obtaining consent), a lactating or pregnant patient, or a patient who may be pregnant (without hysterectomy or ovariectomy) who has no intention to use efficacious contraception defined in this study during the study period and would not agree to receive regular pregnancy tests during the study period
8. A patient who has experienced alcohol abuse or drug abuse within 3 months before obtaining consent, which may disturb the study participation
9. A patient who is in the condition that makes it difficult to administer the study drug
10. A patient with renal dysfunction of eGFR (MDRD calculating formula) <45 mL/min/1.73 m2 prior to starting extension study treatment (Day 0)
11. A patient who indicates a hypersensitivity response to empagliflozin or its excipients, or a patient with lactose-intolerance
12. A patient with severe ketosis, diabetic coma or precoma, severe infection, perioperative status, or serious trauma
13. A patient that the investigator and/or coinvestigator, etc., has judged to be ineligible to this study for other reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events, Adverse drug reactions, and Presence/absence of the use of rescue treatment drugs | until Week 28 (Week 52 of the EMPIRE-01 study)
  Presence/absence of adverse events, adverse drug reactions, and use of rescue treatment drugs

SECONDARY OUTCOMES:
HbA1c change rate at Week 28 (Week 52 of the EMPIRE-01 study) of the treatment from baseline | at Week 28 (Week 52 of the EMPIRE-01 study) of the treatment from baseline
  The HbA1c change rate at Week 28 (52) from baseline is defined as HbA1c change from baseline divided by baseline HbA1c of the EMPIRE-01 study and multiplied by 100.
HbA1c change at Week 28 (Week 52 of the EMPIRE-01 study) of the treatment from baseline | at Week 28 (Week 52 of the EMPIRE-01 study) of the treatment from baseline
  The HbA1c change at Week 28 (52) of the treatment from baseline is defined as the difference in HbA1c levels between Week 28 (52) and baseline of the EMPIRE-01 study.
HbA1c at each time point | at baseline of the EMPIRE-01 study, Week 12 (36), Week 28 (52), or at discontinuation.
  The HbA1c at each time point is defined as the HbA1c levels at baseline of the EMPIRE-01 study, Week 12 (36), Week 28 (52), or at discontinuation.
Fasting plasma glucose (FPG) at each time point | at baseline of the EMPIRE-01 study, Week 12 (36), Week 28 (52), or at discontinuation.
  The FPG at each time point is defined as the FPG levels at baseline of the EMPIRE-01 study, Week 12 (36), Week 28 (52), or at discontinuation.
Fasting plasma glucose (FPG) change at Week 28 (52) of the treatment from baseline | between Week 28 (52) and baseline of the EMPIRE-01 study.
  The FPG change at Week 28 (52) of the treatment from baseline is defined as the difference in the FPG levels between Week 28 (52) and baseline of the EMPIRE-01 study.
Insulin dose at each time point (TDD, TBD) | at baseline of the EMPIRE-01 study, Week 12 (36), Week 28 (52), or at discontinuation.
  The TDD and TBD at each time point are defined as the insulin doses at baseline of the EMPIRE-01 study, Week 12 (36), Week 28 (52), or at discontinuation.
Postprandial glucose for 2 hours over time | for 14 days starting from Week 12 (36)
  Postprandial glucose for 2 hours shall be measured for 14 days starting from Week 12 (36) by using FreeStyle Librae ProTM.

CONTACTS AND LOCATIONS:
Overall Officials: Wataru Ogawa, Study Chair — Kobe University Hospital
Locations (5):
- Japan (5):
  - Kobe University Hospital, Kobe, Hyōgo
  - Tohoku University Hospita, Sendai, Miyagi
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - NIhon University Hospital, Chiyoda-ku, Tokyo
  - Okayama University Hospital, Okayama

IPD SHARING:
Plan to Share IPD: No